CLINICAL TRIAL: NCT06383208
Title: Cardiovascular-Renal Adverse oUtcome rIsk aSsessment systEm for Coronary Heart Disease Complicated With Chronic Kidney Disease Based on Targeted Lipid METabolomics
Brief Title: Cardiovascular-Renal Adverse Prognosis Assessment System for Coronary Heart Disease With Chronic Kidney Disease Based on Metabolomics
Acronym: CRUISE-MET
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Department of Cardiology, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: 2024-ZF-13
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Coronary Heart Disease; Lipid Metabolism Disorders
Keywords: Chronic Kidney Diseases; Coronary Heart Disease; Lipid Metabolism Disorders; Cardiovascular-Renal adverse prognosis; Metabolomics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Disease; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Collect 4 ml of fasting peripheral venous blood from enrolled patients. Fasting should commence at 22:00 the day before blood collection. The blood should be placed in EDTA anticoagulant tubes.
  Within 2 hours after blood collection, plasma should be separated and stored for subsequent lipidomic analysis. This involves centrifuging at 3000 rpm for 10 minutes to separate the plasma. Transfer the upper layer of plasma into 200 ul/1.5 ml EP tubes, then store at -80°C for preservation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lipid metabolomics — Extract 4 milliliters of fasting peripheral venous blood from enrolled patients for targeted lipid metabolism metabolomics research. Utilize a liquid chromatography-tandem mass spectrometry (LC-MS/MS) system to conduct metabolomics analysis on patient blood samples.

SUMMARY:
Coronary heart disease (CHD) combined with chronic kidney disease (CKD) affects a substantial portion of the population and carries a significant disease burden, often leading to poor outcomes. Despite efforts to strictly control traditional risk factors, the efficacy in improving outcomes for patients with both CHD and CKD has been limited. Recent advancements in lipid metabolism research have identified new lipid metabolites associated with the occurrence and prognosis of CHD and CKD. Our preliminary trial has shown that levels of certain lipid metabolites, such as Cer(18:1/16:0), HexCer(18:1/16:0), and PI(18:0/18:1), are notably elevated in patients with CHD and reduced kidney function compared to those with relatively normal kidney function. This suggests that dysregulation of these non-traditional lipid metabolites may contribute to residual risk for adverse outcomes in these patients.

Furthermore, the emerging concept of "cardiovascular-kidney-metabolic syndrome" and the availability of new treatment options highlight the urgent need for a risk stratification tool tailored to modern management strategies and treatment goals to guide preventive measures effectively. To address this, we propose to conduct a prospective cohort study focusing on CHD combined with CKD. This study aims to comprehensively understand the clinical characteristics, diagnosis, treatment status, and cardiovascular-kidney prognosis in these patients. Through advanced metabolomics analysis, we seek to identify lipid metabolism profiles and non-traditional lipid metabolites associated with the progression of coronary artery disease in CHD-CKD patients. Leveraging clinical databases and metabolomics data, we will develop a robust risk prediction model for adverse cardiovascular-kidney outcomes, providing valuable guidance for clinical diagnosis, treatment decisions, and ultimately improving patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Diagnosed with CHD during hospitalization through coronary angiography, including ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation acute coronary syndrome (NST-ACS), stable angina pectoris;
3. Patients with clarified renal function status.;

CKD is defined as meeting one of the following criteria, with a duration of more than 3 months: eGFR < 60 ml/min/1.73 m² or eGFR ≥ 60 ml/min/1.73 m² and urinary albumin-to-creatinine ratio (uACR) ≥ 30 mg/g;

Exclusion Criteria:

1. Pregnancy or lactation;
2. Severe valve disease or severe mechanical complications requiring surgical intervention;
3. Severe psychiatric illness or other reasons that impede follow-up compliance;
4. Severe hematologic disorders or end-stage malignant tumors;
5. Having undergone kidney transplantation or long-term maintenance dialysis;
6. Severe liver disease (Child-Pugh class C);
7. Received acute renal failure dialysis treatment within 12 weeks prior to screening for enrollment;
8. Severe chronic lung disease requiring long-term mechanical ventilation support or awaiting lung transplantation;
9. Life expectancy less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this study will be selected from China-Japan Friendship Hospital
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular adverse events | 12 month follow-up
  Cardiovascular adverse events includes Cardiovascular-related death, non-fatal myocardial infarction, non-fatal stroke, repeat revascularization, rehospitalization for heart failure.
  1. Cardiovascular events related to mortality: This includes 1) cardiovascular death; 2) death caused by stroke; 3) death resulting from cardiovascular surgery; 4) death from other cardiovascular causes.
  2. Cardiovascular death: During the follow-up period, this refers to death directly associated with documented myocardial infarction, heart failure, or arrhythmia. It also includes death events where the cause is unclear and not attributed to any other underlying conditions.
  3. Repeat revascularization is any unplanned repeat revascularization of either a target vessel or non-target vessel or CABG;
Incidence of Renal composite endpoint event | 12 month follow-up
  Renal composite endpoint event includes renal failure, renal-related death, or a decrease in eGFR >40% from baseline (confirmed by a second test 4 weeks later).
  1. Renal failure: End-stage kidney disease (ESKD) or eGFR persistently below 15 ml/min/1.73 m².
  2. End-stage kidney disease: Receiving renal replacement therapy (RRT), including hemodialysis/peritoneal dialysis, for more than 3 months, or undergoing kidney transplantation. Acute kidney injury (AKI) events leading to dialysis and death are also considered end-stage kidney disease (ESKD) events.
  3. Renal-related death: Meeting both of the following criteria: 1) The patient died during the follow-up period; 2) Despite the need for renal replacement therapy (RRT) due to their condition, it was not received；3）No other clear cause of death.

SECONDARY OUTCOMES:
Incidence of All-cause mortality | 12 month follow-up
  All-cause deaths includes cardiac death, vascular death and non-cardiovascular death.
  1. Cardiac death: any death due to proximate cardiac cause (eg, MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  2. Vascular death: caused by noncoronary vascular causes, such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular diseases.
  3. Non-cardiovascular death: any death not covered by the above definitions, such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide, or trauma
Incidence of Repeat revascularization | 12 month follow-up
  Repeat revascularization is any unplanned repeat revascularization of either a target vessel or non-target vessel or CABG.
Incidence of bleeding | 12 month follow-up
  Bleeding Academic Research Consortium (BARC) type 2 to 5 bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Jingang, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided